CLINICAL TRIAL: NCT05112666
Title: Observational Studies in Cancer Associated Thrombosis for Rivaroxaban - United Kingdom Cohort (OSCAR-UK)
Brief Title: A Study to Gather Information About Rivaroxaban in Patients in the United Kingdom Who Have Cancer and Thrombosis (OSCAR-UK)
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 22020
Record Dates: First submitted 2021-10-28; First posted 2021-11-09 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Treatment of Venous Thromboembolism in Cancer Patients
MeSH Terms: interventions — Rivaroxaban; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer patients with VTE: Adults diagnosed with active (primary or metastatic) cancer experiencing a hospitalization or emergency department admission or a primary care visit with an incident venous thromboembolism (VTE), being administered rivaroxaban or other direct-acting oral anticoagulants (DOACs) or a low molecular weight heparin (LMWH) will be included.
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939); Drug: other DOACs; Drug: LMWH

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Retrospective cohort analysis using Clinical Practice Research Datalink (CPRD) GOLD and Aurum Hospital Episode Statistics (HES)-linked datasets in UK.
Drug: other DOACs — Retrospective cohort analysis using CPRD GOLD and Aurum HES-linked datasets in UK.
Drug: LMWH — Retrospective cohort analysis using CPRD GOLD and Aurum HES-linked datasets in UK.

SUMMARY:
Patients with cancer are more likely than those without cancer to develop blood clots (deep vein thrombosis and pulmonary embolism), which are treated using blood thinners (anticoagulants). When clots occur, cancer patients carry a higher risk of recurring clots and more likely to bleed on blood thinning treatments. Therefore, it is critical to use blood thinners that optimize the safety and benefits.

There are two main types of blood thinners that are recommended. The tablets which are direct-acting oral anticoagulants and the injections (low molecular-weight heparin). Clinical trials show the tablets may reduce clot risk but may potentially lead to more frequent bleeding, particularly in those with certain risk factors such as stomach ulcers, previous bleeding problems, certain cancer type.

We aim to examine the effectiveness and safety of the tablets versus the injections for treatment of clots in cancer patients, to better understand these treatments' benefits and risks.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥18 years of age at the time of anticoagulation initiation
* Have active cancer and acute deep vein thrombosis (DVT) and/or pulmonary embolism (PE)
* Treated with rivaroxaban (or any DOAC) or LMWH as their first recorded anticoagulant prescription 7 to 30 days post-acute CAT event diagnosis
* Have been active in the data set for at least 12-months prior to the index event and had at least one provider visit in the 12-months prior to the acute VTE event

Exclusion Criteria:

* Evidence of atrial fibrillation, recent hip/knee replacement (with 90 days of CAT), ongoing VTE treatment, valvular heart disease defined as any rheumatic heart disease, mitral stenosis or mitral valve repair/replacement
* History of inferior vena cava filter before cohort entry
* vitamin K antagonist (VKA) use between cohort entry and index day (initiation of DOAC or LMWH)
* Evidence of any type of therapeutic anticoagulation use during all available look-back period per written prescription or patient self-report
* Initiation of rivaroxaban or other DOACs or LMWH during the study period at non-therapeutic doses (e.g., enoxaparin at a dose other than 1 mg/kg twice daily or 1.5 mg/kg once daily; dalteparin at a dose other than 200 IU/kg of total body weight)
* Pregnancy
* Recording indicative of palliative care before cohort entry
* Any clinically-relevant bleeding-related d hospitalization or VTE recurrence between the initial CAT and the start of observation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with active (primary or metastatic) cancer experiencing a hospitalization or emergency department admission or a primary care visit with an incident VTE, being administered rivaroxaban or other DOACs or a LMWH on or after January 1, 2013.
Sampling Method: Non-Probability Sample
Enrollment: 2601 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
The risk of recurrent VTE at 3-months | Retrospective data analysis from 2013 to 2020
Composite of any major bleeding or clinically-relevant non-major bleeding-related hospitalization at 3-months | Retrospective data analysis from 2013 to 2020
  Per the International Society on Thrombosis and Haemostasis (ISTH) criteria [9, 10] for identification of bleeding-associated hospitalizations.
All-cause mortality at 3-months | Retrospective data analysis from 2013 to 2020

SECONDARY OUTCOMES:
Recurrent VTE at 6- and 12-months post-index VTE | Retrospective data analysis from 2013 to 2020
Composite of any major or clinically-relevant non-major bleeding-related hospitalization at 6- and 12-months post-index VTE | Retrospective data analysis from 2013 to 2020
  Including:
  * Intracranial hemorrhage (ICH)
  * Critical organ bleeding (e.g., intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial bleeding or intramuscular with compartment syndrome)
  * Extracranial bleeding-related hospitalizations (including trauma-related)
Composite of any major bleeding or clinically-relevant non-major bleeding-related hospitalization at 6 and 12-months | Retrospective data analysis from 2013 to 2020
  Per the ISTH criteria [9, 10] for identification of bleeding-associated hospitalizations.
Intracranial hemorrhage (ICH), critical organ bleeding and extracranial bleeding-related hospitalizations as separate outcomes | Retrospective data analysis from 2013 to 2020
All-cause mortality at 6- and 12-months | Retrospective data analysis from 2013 to 2020
Incidence rates of recurrent VTE in rivaroxaban, DOAC and LMWH patients experiencing cancer-associated thrombosis (CAT) regardless of the bleeding risk associated with cancer type | Retrospective data analysis from 2013 to 2020
Any clinically-relevant bleeding-related hospitalization in rivaroxaban, DOAC and LMWH patients experiencing cancer-associated thrombosis (CAT) regardless of the bleeding risk associated with cancer type | Retrospective data analysis from 2013 to 2020
All cause-mortality in rivaroxaban, DOAC and LMWH patients experiencing cancer-associated thrombosis (CAT) regardless of the bleeding risk associated with cancer type | Retrospective data analysis from 2013 to 2020
Duration of anticoagulation treatment | Retrospective data analysis from 2013 to 2020
Discontinuation rates of rivaroxaban, DOAC and LMWH at 3-, 6-, 12-months and all available follow-up | Retrospective data analysis from 2013 to 2020

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.